CLINICAL TRIAL: NCT02069483
Title: Testing Methods of Self-persuasion Involving Cigarette Smoking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Pro00048251
Record Dates: First submitted 2014-02-19; First posted 2014-02-24 (Estimated); Last update posted 2014-09-26 (Estimated); Status verified 2014-09

CONDITIONS: Smoking
Keywords: smoking; smoker; text; smartphone; motivation; quitting; cessation; feedback; messages
MeSH Terms: conditions — Smoking | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Motivational Interviewing (Active Comparator): Subjects will engage in motivational interviewing and come up with messages to motivate quitting during the activity.
  Interventions: Behavioral: Motivational Interviewing
- Tailored Feedback (Active Comparator): Subjects will use reasons for quitting that they provided during the phone baseline for the text messages and audio recordings.
  Interventions: Behavioral: Tailored Feedback

INTERVENTIONS:
Behavioral: Motivational Interviewing — Subjects will engage in motivational interviewing in order to generate motivating messages related to quitting smoking.
  Arms: Motivational Interviewing
Behavioral: Tailored Feedback — Subjects will self-generate reasons they want to quit smoking during the baseline survey and record these reasons during the in-person activity.
  Arms: Tailored Feedback

SUMMARY:
Smokers who are not actively engaged in quitting will participate in a study using self-generated text and audio text messages containing reasons to quit smoking.

DETAILED DESCRIPTION:
Participants must have a smartphone that can accept text messages from an email address and link to a study related website to hear audio recordings, and be willing to receive a text message each weekday for two weeks between 8-9am as part of the study. After completing a phone screener, participants will complete a baseline phone survey. Within two weeks of the baseline survey, participants will come to an in-person session. At that time they will be randomized with equal probability to one of two conditions: 1) Motivational Interviewing (MI), or 2) tailored feedback on reasons for quitting. After undergoing MI or receiving tailored feedback, participants will be asked to generate message that they feel would motivate them to quit. These messages will be both text and audio. After generating and reviewing these messages, participants will then evaluate these messages before ending the laboratory session. Starting two days after their laboratory session, between 8:00am and 9:00am, staff will send participants one of the self-generated text messages with a link to also hear the message; this process will last for two weeks. Within a week of stopping sending messages, participants will be asked to complete a final phone survey to elicit smoking behaviors and provided feedback on the messaging.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* not actively engaged in trying to quit smoking
* must have smoked 100 cigarettes to date
* must smoke at least 1 cigarette per day
* must own smartphone capable of receiving messages from study email
* must agree to receive text messages between 8-9am each weekday for 2 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Number of messages generated during in-person visit | one hour

SECONDARY OUTCOMES:
Quality of messages | before and after completion of the trial, approximately 3 weeks
  Smokers' evaluation of message (e.g., persuasiveness, accuracy/credibility, ease of generating messages).

CONTACTS AND LOCATIONS:
Overall Officials: Isaac Lipkus, PhD, Principal Investigator — Duke University School of Nursing
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States